CLINICAL TRIAL: NCT01075997
Title: The Impact of a Video Cell Phone Reminder System on Glycemic Control in Patients With Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Collaborators: Affinity Networks, Inc. (Industry)
Responsible Party: MAJ Amanda Bell MC,MD, Walter Reed Army Medical Center,
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: WU#07-13025
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Last update posted 2010-02-25 (Estimated); Status verified 2009-06

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A cell phone tips (Experimental): This group will receive a cell phone and cell phone service for 1 year. This group will receive a daily video reminders and tips for the first 6 months of the study. For the second 6 months this group will be seen by their providers at least every 3 months, but the video reminders and and tips will no longer be sent. The group will be instructed on how to use the cell phone. The group will be asked to check blood sugar on a schedule determined by their providers. The group will have blood sugars downloaded from from the glucometer by their providers at every visit and reviewed. The group will have the A1c measured. Also it will have this test repeated about every 3 months. They will continue to have monitored their A1c at 24, 38 and 52 weeks of the study.
  Interventions: Device: cell phone delivered tele-educational
- B no cell phone tips (Active Comparator): This group will receive a cell phone and cell phone service for 1 year. For the second 6 months this group will be seen by their providers at least every 3 months. The group will be instructed on how to use the cell phone.The group will be asked to check blood sugar on a schedule determined by their provider. The groups will have blood sugars downloaded from from the glucometer by their provider at every visit and reviewed. The group will have A1c measured. Also it will have this test repeated about every 3 months. They will continue to have monitored their A1c at 24, 38 and 52 weeks of the study.
  Interventions: Device: cell phone

INTERVENTIONS:
Device: cell phone delivered tele-educational — This group will receive a cell phone and cell phone service for 1 year. This group will receive a daily video reminders and tips for the first 6 months of the study. For the second 6 months this group will be seen by their providers at least every 3 months, but the video reminders and and tips will no longer be sent. The group will be instructed on how to use the cell phone.
  Other Names: A cell phone tips
  Arms: A cell phone tips
Device: cell phone — This group will receive a cell phone and cell phone service for 1 year. For the second 6 months this group will be seen by their providers at least every 3 months. The group will be instructed on how to use the cell phone.The group will be asked to check blood sugar on a schedule determined by your provider. The groups will have blood sugars downloaded from from the glucometer by your provider at every visit and reviewed.
  Other Names: B no cell phone tips
  Arms: B no cell phone tips

SUMMARY:
The purpose of the study is to determine whether having a video cell phone that gives daily reminders over a 6-month period to check blood surgery and take your diabetes medications can improve your diabetes control during that time and if that benefit lasts for up to 1 year.

DETAILED DESCRIPTION:
The purpose of this study is to determine if a cell phone video reminder system will improve compliance and glycemic control in patients with diabetes mellitus when compared with standard of care. We plan to partner with Affinity Network, Inc., a local minority-owned small business, to provide broadband-enabled cell phone service to patients with diabetes mellitus. Their IntelaCare™ system will host the content and transmit it to the phones on a personalized schedule. This will be a prospective, randomized, controlled trial comparing patients with diabetes mellitus who receive daily video reminders via cell phone to take their medications and check their blood glucose with patients who are just given a cell phone without daily reminders. The primary endpoint will be improvement of glycemic control as measured by glycosylated hemoglobin (A1c). The secondary endpoints will compare mean daily glucose levels, the number of both hypoglycemic and hyperglycemic events, the amount of time spent in target blood glucose, and the perceived level of diabetes-related stress between the two groups. Patients in both groups will receive a broad-band enabled cell phone and cell phone service for the duration of the study. Patients will be randomized into a "cell phone" group (group A) and a "cell phone plus reminder" group (group B). They will be seen by their provider at least quarterly (or more often as clinically appropriate). Blood glucose readings will be downloaded from patients' glucometers at every provider visit (at least quarterly). Group B will receive a daily 15-second video from their provider reminding them to take their medication and to test their blood sugar and an educational "tip-of-the day." These reminders will be personalized and recorded by their provider. During the second 6 months, the patients will be followed by their provider at least quarterly. Improvement in glycemic control will be determined by quarterly measurements of A1c and the mean and standard deviation of blood glucose. In addition, the number of home blood glucose tests performed on a weekly basis will be compared. Compliance with medication will be determined by pharmacy refill records and pill counts. Quality-of-life will be measures using 2 validated instruments at 0, 26 and 52 weeks - the Problem Areas in Diabetes (PAID), which is a diabetes-related quality of life questionnaire and the SF-8, which is a general quality of life questionnaire for people with chronic disease.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or greater
* A1c greater than 8%
* ability to use a cell phone and glucose meter
* ability to understand English
* on oral therapy and/or insulin

Exclusion Criteria:

* under age 18
* non-English speaking
* females who are pregnant, lactating, planning to become pregnant, or without a safe contraceptive method
* A1c less than 8%
* use of glucocorticoids, amphetamines, anabolic, or weight-reducing agents during the course of the study

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2007-11; Primary Completion 2010-07 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will be improvement of glycemic control as measured by glycosylated hemoglobin (A1c). | week 0, week 12, week 26, week 38, week 52

SECONDARY OUTCOMES:
To compare mean blood glucose levels,the number of hypo- and hyperglycemic events,the duration of time spent in target blood glucose range,the perceived level of diabetes-related stress and the perceived effect of diabetes on quality of life. | week 0, week 12, week 26, week 38, week 52

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Bell, MD, Principal Investigator — WRAMC
Locations (1):
- Walter Reed Army Hospital Center, Washington D.C., District of Columbia, United States